CLINICAL TRIAL: NCT02182492
Title: Comparison of Different Efficacy of Macrolide and Glucocorticoid in the Treatment of Chronic Rhinosinusitis Patients After Endoscopic Sinus Surgery
Brief Title: Efficacy of Macrolide and Glucocorticoid in the Treatment of Chronic Rhinosinusitis After Endoscopic Sinus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zheng Liu (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor-Investigator, Zheng Liu, Professor of Otolaryngology-Head & Neck Surgery Vice Director Department of ENT Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENTDrug-001
Record Dates: First submitted 2014-06-30; First posted 2014-07-08 (Estimated); Results first posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Chronic Rhinosinusitis; Endoscopic Sinus Surgery
MeSH Terms: interventions — Clarithromycin; Glucocorticoids; Fluticasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glucocorticoid (Experimental): Fluticasone propionate nasal spray
  Interventions: Drug: Glucocorticoid
- Clarithromycin (Experimental): Clarithromycin tablet
  Interventions: Drug: Clarithromycin

INTERVENTIONS:
Drug: Clarithromycin — Clarithromycin 250 mg tablet once daily for 3 months
  Other Names: KLACID
  Arms: Clarithromycin
Drug: Glucocorticoid — Fluticasone propionate nasal spray 200 μg/d for 3 months
  Other Names: FLIXONASE
  Arms: Glucocorticoid

SUMMARY:
Endoscopic sinus surgery (ESS) is widely considered to be the gold standard in the surgical management of chronic rhinosinusitis (CRS) that has failed maximal medical therapy. Nevertheless, the postoperation medical therapy was considered as a crucial procedure for the success of ESS. Both glucocorticoids and macrolide antibiotics have been recommended for the treatment of CRS, but their effect as postoperation medical therapies of ESS need more clinical data to clarify.

The purpose of this prospective, randomized,study is to determine the effect of glucocorticoids and macrolide antibiotics for the postoperation medical therapy of ESS in different subtypes of CRS.

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS) is a multifactorial inflammatory disorder that causes various symptoms including nasal obstruction, rhinorrhea, olfactory dysfunction, facial pain, and headache . Endoscopic sinus surgery (ESS) is usually recommended for patients who do not response well to conservative treatments. Although surgery is effective to alleviate symptoms and improve the quality of life of CRS patients, a followed long-term postoperative medical treatment is indispensable. Current European and American guidelines recommend glucocorticoids and antibiotics as the primary pharmacotherapeutic approaches for CRS before and after ESS. However, there are a number of CRS patients not responding well to glucocorticoid treatment and conflicting results exist regarding the efficacy of long-term, low-dose macrolide treatment. One potential reason is that CRS is a heterogeneous group of disorders unified by similar clinical presentations and its phenotypes and/or endotypes may be important factors determining the efficacy of treatments.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the CRS diagnostic criteria including CRSsNP and CRSwNP based on the EP3OS definition
* Age ≥16 and ≤70 years
* Chinese of either sex
* Failure to conventional medical therapies according to EP3OS recommendation

Exclusion Criteria:

* Pregnant or breast-feeding women
* Cystic fibrosis
* Congenital ciliary dyskinesia
* Sinonasal fungal disease
* Systemic vasculitis
* Granulomatous disease
* Tumor
* Immunodeficiency
* Allergic to clarithromycin or topical corticosteroid
* With an upper respiratory tract infection within 4 weeks of entering the study
* With serious metabolic, cardiovascular, autoimmune, neurology, blood, digestive, cerebrovascular, respiratory system disease, or any disease interfering with the evaluation of results or affecting subjects' safety such as glaucoma and tuberculosis
* With emotional or mental problems
* Have received immunotherapy within the previous 3 months
* Have had a history of local or systemic medications, such as glucocorticoids and macrolides within 4 weeks
* Have had an acute asthmatic within the 4 weeks before entering the study

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Liu, Doctor, Study Director — Professor of Otolaryngology-Head & Neck Surgery Vice Director Department of ENT Tongji Hospital Tongji Medical College Huazhong University of Science and Technology
Locations (1):
- Department of ENT, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients meeting the Chronic rhinosinusitis (CRS) diagnostic criteria outlined in the European Position Paper on Rhinosinusitis and Nasal polyps (EP3OS) definition were enrolled. Three subtypes CRS included: CRS without nasal polyps (CRSsNP); non-eosinophilic CRS with nasal polyps (Non-Eos CRSwNP); eosinophilic CRS with nasal polyps (Eos CRSwNP).
Period: Overall Study
Arm/Group | Glucocorticoid | Clarithromycin
Started | 93 (CRSsNP: 28; Non-Eos CRSwNP: 34; Eos CRSwNP: 31) | 94 (CRSsNP: 30; Non-Eos CRSwNP: 32; Eos CRSwNP: 32)
Completed | 86 (CRSsNP: 27; Non-Eos CRSwNP: 31; Eos CRSwNP: 28) | 86 (CRSsNP: 29; Non-Eos CRSwNP: 28; Eos CRSwNP: 29)
Not Completed | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glucocorticoid | Clarithromycin | Total
Number analyzed (Participants) | 93 | 94 | 187
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 5 | 12
  Between 18 and 65 years | 84 | 86 | 170
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (12.6) | 39.9 (14.2) | 40.2 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 42 | 80
  Male | 55 | 52 | 107
Region of Enrollment [Number; unit: participants]
  China | 93 | 94 | 187

OUTCOME MEASURES:

1. Primary Outcome: Total Subjective Symptoms Visual Analog Scores (VAS)
Description: The treatment will begin one week after ESS. Symptoms visual analog scores (VAS) were recorded just before ESS and at 1-, 3-, 6- and 12-month follow-up visit. All of the patients were assessed by using symptom questionnaire after enrollment and at follow-up visits. Subjective symptoms were scored by patients on a VAS of 0-10, with 0 being "no complaint whatsoever" and 10 being "the worst imaginable complaint."Five major symptoms were focused on: nasal obstruction, rhinorrhea, loss of sense of smell, facial pain or pressure, and headache. Total VAS score was calculated based on the sum of VAS scores of these five symptom domains. Total subjective symptoms VAS range: 0~50, with higher scores indicating greater severity of symptoms.
Time Frame: Scores will be recorded just before ESS and at 1-, 3-, 6- and 12-month follow-up visit.
Population: A total of 187 patients met the study eligibility criteria. Seven patients in fluticasone propionate group and 8 patients in clarithromycin group dropped out because of nonadherence.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Glucocorticoid | Clarithromycin
Number analyzed (Participants) | 86 | 86
score on a scale
  Baseline | 20.4 (8.1) | 20.7 (7.8)
  1-month | 9.7 (5.2) | 8.9 (5.0)
  3-month | 7.0 (4.2) | 5.8 (4.3)
  6-month | 5.9 (4.5) | 4.7 (4.2)
  12-month | 5.6 (5.3) | 4.8 (5.0)

2. Secondary Outcome: Total Nasal Endoscopic Scores
Description: Nasal endoscopic evaluation was performed by the senior investigator who remained blinded to the treatment, including poly size: 0, absence of polyps; 1, polyps in middle meatus only; 2, polyps beyond middle meatus but not blocking the nose completely; and 3, polyps completely obstructing the nose; discharge: 0, no discharge; 1, clear thin discharge; 2, thick purulent discharge; edema: 0, no edema; 1, mild edema; 2, severe edema; crusting: 0, no crusting; 1, mild crusting; 2, severe crusting; scarring: 0, no scarring; 1, mild scarring; 2, severe scarring). Each side was graded separately, and the scores from both sides were added to determine the overall scores for a particular domain. The total endoscopy score was calculated based on the sum of scores of these endoscopic domains. Endoscopic scores were also recorded before ESS (baseline) and at 1-, 3-, 6- and 12-month follow-up visits. Total endoscopy score range: 0~22, with higher scores indicating greater severity.
Time Frame: Scores will be recorded just before ESS and at 1-, 3-, 6- and 12-month follow-up visit.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Glucocorticoid | Clarithromycin
Number analyzed (Participants) | 86 | 86
score on a scale
  Baseline | 8.2 (2.9) | 7.6 (2.9)
  1-month | 5.3 (2.3) | 4.7 (2.2)
  3-month | 3.7 (2.8) | 3 (2.4)
  6-month | 3.1 (2.6) | 2.1 (2.2)
  12-month | 2.7 (2.6) | 2.1 (2.4)

3. Other Pre Specified Outcome: Measurement of Protein Levels of Inflammatory Molecules in Tissues
Time Frame: Polyp tissues from CRSwNP patients and diseased sinus mucosa from CRSsNP patients will be collected during surgery.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Glucocorticoid | Clarithromycin
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/94
Other Adverse Events (participants affected / at risk) | 5/93 | 5/94
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Glucocorticoid (N=93) | Clarithromycin (N=94)
Mild nasal bleeding (Surgical and medical procedures) | 3 | 2
Mild diarrhea (Surgical and medical procedures) | 1 | 2
Headache (Surgical and medical procedures) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes